CLINICAL TRIAL: NCT00915109
Title: Gait Stability of People With Lower-limb Amputations
Status: Completed | Type: Observational
Sponsor: Kim Parker (Other)
Responsible Party: Sponsor-Investigator, Kim Parker, Rehabilitation Engineer, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: CDHA-RS-2010-026
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Gait; Balance
Keywords: amputees; lower limb

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- vascular: People with a unilateral below-knee amputations due to a vascular reason
- nonvascular: People with a below-knee amputation due to nonvascular reasons
- Control: People with no gait impairments.

SUMMARY:
The purpose of this study is to evaluate whether there are quantifiable differences in walking stability, as measured by the acceleration of the trunk or the variation in step length, between people with unilateral below-knee amputations from vascular reasons or from trauma reasons.

ELIGIBILITY:
Inclusion Criteria:

* be over the age of 18;
* be able to walk comfortably for a minimum of two (2) minutes;
* be willing to take part in the study, including signing the consent after carefully reading it;
* be able to read and understand English and follow verbal and visual instructions;
* are competent to give informed consent or have a proxy with power of attorney.
* have an unilateral, transtibial amputation;
* been fitted with a prosthesis for over six weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prosthetic outpatient clinic of one rehabilitation centre
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada